CLINICAL TRIAL: NCT02797678
Title: A Double-Blind Placebo-Controlled Multi-Site Randomized Cross-Over Study of the Feasibility, Effectiveness and Efficacy of the PowerSleep Device
Brief Title: Feasibility, Effectiveness and Efficacy of the PowerSleep Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CAI-16025-PSPIL-LO
Record Dates: First submitted 2016-05-20; First posted 2016-06-13 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Sleep; Sleep Disorders Not Due to A Substance or Known Physiological Condition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Powersleep Stim, PowerSleep Sham (Experimental): Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night for one week. Participants will then be crossed over and will wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers for one week
  Interventions: Device: Powersleep; Device: Sham Powersleep
- Powersleep Sham, PowerSleep Stim (Sham Comparator): Participants wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers for one week. Participants will then wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night for one week.
  Interventions: Device: Powersleep; Device: Sham Powersleep

INTERVENTIONS:
Device: Powersleep — Participants will receive 5 nights of stimulation
Device: Sham Powersleep — Participants will receive 5 nights of no stimulation

SUMMARY:
The purpose of this study is test the effectiveness of the PowerSleep auditory stimulation device on sleep quality and daytime functioning in individuals who have insufficient sleep.

The PowerSleep device is a non-invasive portable device designed to increase deep sleep, potentially reducing daytime sleepiness related to insufficient sleep. The device is meant to be worn while a person is sleeping. The device delivers soft audio tones (below 65dB (decibels)/ normal speaking voice) via headphones periodically throughout the night and records the electrical activity of the brain (electroencephalogram (EEG)). The device consists of a headband with 4 sensors on the forehead, one sensor behind the right ear, headphones covered by speaker foam over each ear, and a cable which connects the headband to an upper arm band. The armband contains the device electronics. The headband and the armband are connected via adjustable Velcro closure. This device has not been released for sale and is considered investigational.

The study includes approximately 30 people from four study sites. It is anticipated that a total of up to 10 people will complete the study at this site. This study is designed to last up to 6 weeks.

DETAILED DESCRIPTION:
PowerSleep is a non-invasive portable light weight device designed to stimulate deep slow-wave sleep and thereby reduce daytime sleepiness associated with insufficient sleep or poor perceived sleep quality. The concept is to stimulate deep sleep also known as (Slow-Wave Sleep [SWS]), to compensate for insufficient sleep duration by increasing sleep intensity or to improve sleep quality by increasing sleep intensity. Sleep intensity can be objectively assessed by Slow-Wave Activity (SWA). In normal individuals, a reduction in amounts of SWA consistently results in reduced alertness with impaired performance due to cognitive and memory deficits.

The PowerSleep device delivers acoustic stimuli that are calibrated to stimulate SWA without awakening the user. The PowerSleep device is wearable and non-invasive, consisting of a headband with 4 integrated electrodes and headphones covered by speaker foam over each ear. The headband is connected via a tether cable to an upper arm band which houses the EEG amplifier and electronics of the device. Both the headband and the arm band are adjusted via a Velcro strap. The device also includes a right mastoid electrode. The device monitors and records EEG throughout the night, and is capable of on-line identification of sleep stages and continuous EEG analysis. The armband contains the device electronics. EEG data collected by the PowerSleep device can be transferred to the computer by a technician after home use and used to assess sleep quality. Soft audio tones will be administered via the speakers during deep sleep throughout the night.

Participants may be pre-screened over the phone to determine eligibility. A screening script will include a general review of key inclusion and exclusion criteria, and questionnaires to assess the risk of an undiagnosed sleep disorder. Participants that meet all eligibility criteria will be asked to come into the lab for a screening daytime visit (Visit 1) involving a detailed presentation of the study and an interview to verify eligibility and work schedules.

Participants who are interested and eligible will be consented. Participants will scheduled for up to 6 daytime visits, 2 overnight lab visits, and provided with information on use of the actigraph and PowerSleep device at home. At Daytime Visit 2, participant qualification will be assessed based on the PowerSleep device data. Qualifying participants will be randomized and receive a PowerSleep device for home use.

Participants will use the PowerSleep device with active and sham study arm for one work week each, with a washout period in between. At the end of each study arm work week, the participants will report to the lab for an overnight stay followed by daytime in- lab testing to complete daytime function assessments and questionnaires. Compliance data from the PowerSleep device will be reviewed at each visit, and only qualifying participants will continue in the study.

Daytime Visit 1 Procedures (Up to 2 hours):

Initial evaluation and anthropometric measurements:

Participants will be asked to report to the sleep lab for a daytime visit. A detailed interview will be performed verifying eligibility criteria, and review of work and non-work schedules. After a full explanation of the protocol and after all the participants' questions have been answered, participants will be asked to sign the consent form.

Participants will be asked to fill out the baseline questionnaires, medical history, review of systems, and current medications.

Participants will have height, weight, waist to hip ratio, neck circumference, heart rate (after being seated for approximately 5 minutes), temperature, respiratory rate and blood pressure (systolic and diastolic after being seated for approximately 5 minutes) recorded.

Participants will be trained in the use of the sleep logs, actigraphy and be fitted and trained on the device use for baseline night data collection.

Actigraphy screening:

Participants will be asked to wear an actigraph and complete a daily sleep logs for up to 7 days (including at least 3 workdays) including monitoring a sleep schedule. Participants will receive instructions from the study staff on how to wear the actigraph and will be asked to keep to a regular sleep schedule.

Baseline Night training:

Participants will be asked to wear the PowerSleep device at home for one night. During the Daytime Visit, participants will be fitted with PowerSleep device and trained on its use for data collection on the baseline night.

Participants will receive a phone call from the study staff as a reminder to wear the device on the appropriate night for the baseline data collection.

After the initial screening, participants will be asked to report to the lab (Daytime Visit 2) for equipment and sleep log return, and download and review of study data.

Daytime Visit 2 Procedures (2 hours):

Participants will return to the sleep lab (within 1 week of daytime visit 1, ±2 days) with the actigraph, sleep diary and PowerSleep device for review by the study staff.

Actigraphy review:

The sleep log and actigraph data will be reviewed by a trained technologist prior to randomization.

Baseline Night review:

The PowerSleep device data will be downloaded and reviewed. Qualifying participants will be asked to continue wearing the actigraph and completing the sleep diary throughout the study.

Participants will be asked questions related to the comfort, the ease of use and overall device use after the baseline night

Device home use:

Once eligibility has been confirmed, participants will be re-trained on the study device take home use. Participants will be asked to use the device during 5 consecutive workday nights (Monday - Thursday) at home and Friday night overnight in the lab in order to be eligible for continued study participation. In addition, at least 4 hours of device use per night is required for study continuation. Participants will be instructed that the device must be used nightly; and imperative to be used prior to morning recall assessment cognitive measures (Monday nights (initial night) of each work week use and Friday nights during the overnight in lab visit).

Participants will be randomly assigned to active or sham treatment during the first work week in a 1:1 ratio. Participants and study staff will be blinded to the treatment during each work week.

Active treatment: Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night.

Sham treatment: Participants wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers.

Daytime assessments:

Participants will also be trained on daytime assessments and asked to complete a battery at home in the morning.

Overnight in-lab visit (8-12 hours) followed by Daytime in-lab testing (8 hours): On Friday evening participants will be asked to return to the sleep lab for an overnight visit. Participants will be asked to report to the lab 1.5 to 2 hours before bedtime with all study materials including the logs, questionnaires, device and laptop. Participants will be asked to go to bed and awaken at the same time as a regular work-night sleep schedule. Participants will be asked to continue to wear the PowerSleep device during this overnight visit.

On the morning of the day following the overnight in lab visit work week 1, participants will remain in the lab and undergo the following assessments:

* Review of any reported changes in medical condition since previous visit
* Collect sleep logs
* Collect PowerSleep device
* Data download from actigraph and study device with verification of device compliance
* Collect daily home assessments of daytime function
* Three consecutive blood pressure measurements at 5 min intervals while sitting
* Complete questionnaires
* Complete 3 minute Psychomotor Vigilance Task (PVT)
* active vs sham
* Complete morning recall of Paired Associated Learning (PAL) task
* A single fasting blood draw for glucose and insulin
* Breakfast- participants can have one (1) 6 ounce cup of coffee or caffeine equivalent. Coffee or equivalent is only for those who routinely drink caffeine in the morning.
* 4- nap Multiple Sleep Latency Test (beginning standardly 2 hours post wake-up): each nap is followed by a battery of assessments which includes questionnaires and a the 3 min PVT.

Participants will enter into a washout period of 1 to 2 weeks at which time participants will continue to wear the actigraph and complete sleep logs and will not use the Powersleep device.

Daytime Visit 4 (1 hour):

Participants will report to the lab and receive the PowerSleep device for the 2nd work week use period. Participants will be re-trained on the home use of the device and will be asked to use the device during 5 consecutive workday nights. Sleep logs will be collected and reviewed with actigraph data.

Participants will be crossed over to other study arm at the time of this visit.

Overnight in-lab visit (8-12 hours) followed by Daytime in-lab testing (8 hours):

This is a repeat of the above day-time in lab testing.

Participants will be asked to continue wearing actigraph over the weekend for the purposes of collecting data related to recovery sleep at end of study.

Daytime Visit 6 (30 minutes) Participants will be asked to return to the lab for a quick visit to return actigraph and data download capturing recovery sleep.

Participants will be asked questions related to the comfort, the ease of use and overall device use after two weeks of home use.

Statistics:

Descriptive statistics will be presented for all variables of interest. Continuous data will be summarized by mean, standard deviation, median, minimum, and maximum values. Categorical data will be presented as frequencies and percentages. Endpoints will be compared between the active and sham conditions as paired samples. Continuous endpoints that are not normally distributed may undergo appropriate transformation to fit the assumptions of a paired t-test. Otherwise, the nonparametric Wilcoxon Signed Ranks test will be used. Categorical endpoints will be examined with the McNemar Test. All tests will be conducted at a significance level of p < 0.05.

Data quality will be assessed by the blinded personnel scoring the PSGs (Polysomnography) and device data. Criteria will be defined regarding whether the data sets are scorable and of sufficient duration to be included in the statistical analysis. These criteria will be consistently applied across all participant records and described in any study publications or reports.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to admission
* Able to read, write and speak English
* Adult volunteers aged 21-50 working full time; 5 consecutive days (M-F)
* Self-reported regular sleep schedule
* Self-reported sleep duration of > 5hrs. and ≤ 6.5hrs. (verified by 3 work days of ambulatory sleep monitoring with wrist actigraphy and daily logs)
* Self-reported sleep latency > 30 minutes no more than once / wk. (time to fall asleep)
* Self-reported wake after sleep onset ≤ 30 minutes
* Participants who regularly use an alarm clock during the work week and who self-report:

  i. Regular time in bed (TIB) on work days of ≤7 hours ii. Regular increase in sleep duration by ≥ 1 hour during non-work days as compared to work days, either by nocturnal bedtime extension of via a daytime nap

Exclusion Criteria:

* Participation in another interventional study in the past 30 days.
* Major controlled or uncontrolled medical condition such as congestive heart failure, neuromuscular disease, renal failure, cancer, Chronic Obstructive Pulmonary Disease (COPD), respiratory failure or insufficiency, or patients requiring oxygen therapy (as determined by self-report and reviewed by the study PI.)
* Currently working night shift or rotating shift.
* Current use or use of within the past month of a prescription or over-the-counter sleep medication or stimulant; use of psychoactive medication (based on self-report and review with a study clinician) Refer to table below for examples.
* Pregnancy
* Body Mass Index > 40 kg/m2
* Prior diagnosis of any sleep disorder including

  1. Obstructive Sleep Apnea (AHI ≥15 events/hour) - from ambulatory or in lab polysomnography
  2. Restless legs syndrome, or periodic limb movement disorder
  3. Insomnia
  4. Parasomnia
* High Risk of OSA (Obstructive Sleep Apnea) based on STOP-BANG Questionnaire ("yes" on at least 3 of 7 questions)
* High Risk of Restless Legs Syndrome (RLS) based on Cambridge-Hopkins Screening questionnaire
* Excessive alcohol intake (self-report > 14 drinks / wk.)
* Self-report of binge alcohol consumption ( >5 drinks) on any one day during the week prior to the randomization, during the device use period, and during the wash-out period
* Excessive caffeine consumption (> 500mg/day combining all caffeinated drinks regularly absorbed during workdays.) Caffeine intake must be regular and maintained throughout study and on testing days (available at test sites)
* Individuals who self-report a history of recurrent seizures or epilepsy or have a history of medical conditions that could increase the chance of seizures (e.g. stroke, aneurysm, brain surgery, structural brain lesion).
* Individuals who self-report severe contact dermatitis.
* Individuals who self-report moderate hearing loss.
* Inability to achieve appropriate headband fit.
* Planned air travel or travel across more than one time zone one month prior to and or during the anticipated period of the study with PowerSleep device use

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Rosenberg, PhD, Principal Investigator — NeuroTrials Research, Inc.
Locations (4):
- United States (4):
  - NeuroTrials Research Inc, Atlanta, Georgia
  - St. Lukes Hospital, Chesterfield, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Screening Phase: This is all participants that signed consent for this study.
- PowerSleep Stim, PowerSleep Sham: This arm are participants that were randomized to PowerSleep Stim mode first and then PowerSleep Sham.
- PowerSleep Sham, PowerSleep Stim: This arm are participants that were randomized to PowerSleep Sham first, and then PowerSleep Stim.
- PowerSleep Stim - Extension Study: Those participants that completed the primary trial, participated in an extension study.
Period: Screening Phase
Arm/Group | Screening Phase | PowerSleep Stim, PowerSleep Sham | PowerSleep Sham, PowerSleep Stim | PowerSleep Stim - Extension Study
Started | 62 | 0 | 0 | 0
Completed | 37 | 0 | 0 | 0
Not Completed | 25 | 0 | 0 | 0
Not completed — Meeting Inclusion/Exclusion criteria | 25 | 0 | 0 | 0
Period: First Intervention (5 Nights)
Arm/Group | Screening Phase | PowerSleep Stim, PowerSleep Sham | PowerSleep Sham, PowerSleep Stim | PowerSleep Stim - Extension Study
Started | 0 | 20 | 17 | 0
Completed | 0 | 19 | 17 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — study/device use non-compliance | 0 | 1 | 0 | 0
Period: Washout
Arm/Group | Screening Phase | PowerSleep Stim, PowerSleep Sham | PowerSleep Sham, PowerSleep Stim | PowerSleep Stim - Extension Study
Started | 0 | 19 | 17 | 0
Completed | 0 | 19 | 17 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (5 Nights)
Arm/Group | Screening Phase | PowerSleep Stim, PowerSleep Sham | PowerSleep Sham, PowerSleep Stim | PowerSleep Stim - Extension Study
Started | 0 | 19 | 17 | 0
Completed | 0 | 19 | 16 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — study/device use non-compliance | 0 | 0 | 1 | 0
Period: Sub-Study
Arm/Group | Screening Phase | PowerSleep Stim, PowerSleep Sham | PowerSleep Sham, PowerSleep Stim | PowerSleep Stim - Extension Study
Started | 0 | 0 | 0 | 9
Completed | 0 | 0 | 0 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants consented.
Groups:
- All Study Participants: All participants that were consented for this study are including in the baseline measures.
Arm/Group | All Study Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 37
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 62
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Slow Wave Activity Detected by the Powersleep Device With and Without Stimulation
Description: Slow wave activity levels will be compared analyzed by using the PowerSleep Device with stimulation and without stimulation (sham).
  For the analysis of SWA, six-second-long NREM epochs were considered. Every 30 s-long window was subdivided into five epochs and the sleep stage of the window was assigned to every epoch.
  The SWA of each epoch was estimated from the epoch's power spectrum density (PSD) by integrating over the frequency range spanning from 0.5 to 4 Hz.
  The PSD per epoch was estimated according to the Welch method with a four- second long Hanning window (ensuring 0.25 Hz frequency resolution), a two-second-long overlap, and 1024 points to calculate the Fourier transform.
  Since μ-arousal events have spike-like temporal characteristics that manifest as high values in the spectral domain, epochs containing annotated-arousals were discarded from SWA analysis. The average SWA was calculated by taking the average slow-wave activity over all considered NREM epochs
Time Frame: 10 nights
Population: 7 completed participants were excluded from the final analysis for the following reasons: 3 - non-scorable data - signal interference 3 - did not cross over
  1 - did not meet inclusion/exclusion criteria
Measure: Mean (Standard Deviation); unit: microvolts^2
Groups:
- Powersleep: Participants will wear the PowerSleep device with soft audio tones (below 65dB to prevent arousals from sleep) administered via the speakers during deep sleep throughout the night.
  Powersleep: Participants will receive 5 nights of stimulation
- Sham Powersleep: Participants wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers.
  Sham Powersleep: Participants will receive 5 nights of no stimulation
Arm/Group | Powersleep | Sham Powersleep
Number analyzed (Participants) | 28 | 28
microvolts^2 | 1367.9 (491.6) | 1291.3 (431.9)
Statistical Analysis 1: Comparison: Powersleep vs Sham Powersleep; Test type: Superiority; p = 0.061, paired t-test

2. Secondary Outcome: Changes in Vigilance Scores as Measured by the Psychomotor Vigilance Task (PVT)
Description: To measure trends of vigilance of one work week (4 nights of home use and one night in the sleep lab) with active PowerSleep (delivering audio tones) as compared to a one work week (4 nights of home use and one night in the sleep lab) of sham (delivering no audio tones).
  The measure of vigilance scored was average reaction time in milliseconds.
Time Frame: 10 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Powersleep Stim: Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night.
- Powersleep Sham: Sham Powersleep: Participants will receive 5 nights of no stimulation
Arm/Group | Powersleep Stim | Powersleep Sham
Number analyzed (Participants) | 28 | 28
milliseconds | 251.4 (31.47) | 252.1 (32.79)

3. Secondary Outcome: Changes in Memory Scores as Measured by the Paired-Associate-Learning (PAL)
Description: Participants performed a learning activity of an 80 word pair list the night of the in-lab visit and then completed a recall in the morning following the overnight in the sleep lab. The results listed below are the mean and standard deviation of the PowerSleep treatment week compared to the Sham treatment week.
Time Frame: 2 nights
Population: Only 22 participants completed the PAL the morning after the overnight in the sleep lab. 6 participants did not complete the PAL on both nights.
Measure: Mean (Standard Deviation); unit: words
Groups:
- Powersleep: Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night.
Arm/Group | Powersleep | Sham Powersleep
Number analyzed (Participants) | 22 | 22
words | 35.5 (18.23) | 33.86 (16.99)

4. Primary Outcome: Amount of Cumulative Slow Wave Activity Detected by the Powersleep Device With and Without Stimulation
Description: For the analysis of SWA, six-second-long NREM epochs were considered. Every 30 s-long window was subdivided into five epochs and the sleep stage of the window was assigned to every epoch.
  In our research, both SWA and CSWA are evaluated as relative values having as reference the average SWA and CSWA over sham sleep sessions. CSWA is the integral of SWA which is why the unit of CSWA is microvolt^2×minute.
Time Frame: 10 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microvolts^2x minute
Arm/Group | Powersleep | Sham Powersleep
Number analyzed (Participants) | 28 | 28
microvolts^2x minute | 1333663.5 (583242.2) | 1462267.3 (852742.1)
Statistical Analysis 1: Comparison: Powersleep vs Sham Powersleep; Test type: Superiority; p = 0.301, paired t-test

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Screening - Non Intervention: SThe adverse events are reported on all participants that entered screening for the study until randomization visit
- PowerSleep Stim: All participants that received the PowerSleep Stim week.
- Washout: All participants that had a washout period of one to two weeks before crossing over into the other arm of the trial.
- Powersleep Sham: All participants that received the PowerSleep Sham week
- Sub-study: Completed participants were asked to participate in a sub-study with a new device configuration. Participants completed 5 nights of use.
Arm/Group | Screening - Non Intervention | PowerSleep Stim | Washout | Powersleep Sham | Sub-study
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/35 | 0/36 | 0/36 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/35 | 0/36 | 0/36 | 0/9
Other Adverse Events (participants affected / at risk) | 7/62 | 6/35 | 2/36 | 5/36 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screening - Non Intervention (N=62) | PowerSleep Stim (N=35) | Washout (N=36) | Powersleep Sham (N=36) | Sub-study (N=9)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (2) | 2 (2) | 0 (0)
Difficulty Sleeping (General disorders) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
A limitation of this study is the use of generic algorithm parameters that were applied to all participants and the analysis of the effects was performed on the signal recorded by the device in the absence of simultaneously recording PSG data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No